CLINICAL TRIAL: NCT01607918
Title: Comparison of the Efficacy of Clarithromycin-based Triple Therapy for 14 Days Versus Sequential Therapy for 10 Days in the First Line Therapy for Helicobacter Pylori Infection- A Multicenter Randomized Comparative Trial
Brief Title: Clarithromycin-based Triple Therapy for 14 Days Versus Sequential Therapy 10 Days in the First Line Therapy
Acronym: THC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Doctor and Principle Investigator, Department of Gastroenterology, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201110019MD
Record Dates: First submitted 2012-02-16; First posted 2012-05-30 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Eradication Rates of the Two Regimens
Keywords: H pylori, eradication
MeSH Terms: interventions — Lansoprazole; Amoxicillin; Clarithromycin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequential therapy 10 days (Experimental): Sequential therapy
  Interventions: Drug: D1-D5: (lansoprazole + amoxicillin ) D6-D10: (lansoprazole+clarithromycin +metronidazole)
- Triple therapy 14 days (Active Comparator): Triple therapy
  Interventions: Drug: D1-D14: (lansoprazole + clarithromycin + amoxicillin)

INTERVENTIONS:
Drug: D1-D5: (lansoprazole + amoxicillin ) D6-D10: (lansoprazole+clarithromycin +metronidazole) — D1-D5: (lansoprazole 30mg + amoxicillin 1gm) bid D6-D10: (lansoprazole 30mg+clarithromycin 500mg+metronidazole 500mg) bid
  Other Names: Takepron; Amoxicillin; Klaricid; Flagyl
  Arms: Sequential therapy 10 days
Drug: D1-D14: (lansoprazole + clarithromycin + amoxicillin) — D1-D14: (lansoprazole 30mg + clarithromycin 500mg + amoxicillin 1gm) bid
  Other Names: Takepron; Klaricid; Amoxicillin
  Arms: Triple therapy 14 days

SUMMARY:
The investigators aimed to compare the eradication rates of sequential therapy for 10 days versus triple therapy for 14 days

ELIGIBILITY:
Inclusion Criteria:

* Patients are aged greater than 20 years who have H. pylori infection without prior eradication therapy and are willing to receive the sequential therapy will be eligible for enrollment.
* Written informed consents will be obtained from all patients prior to enrollment.

Exclusion Criteria:

Patients will be excluded from the study if any one of the following criteria is present:

* children and teenagers aged less than 20 years,
* history of gastrectomy,
* gastric malignancy, including adenocarcinoma and lymphoma,
* previous allergic reaction to antibiotics (amoxicillin, clarithromycin, levofloxacin, metronidazole) and prompt pump inhibitors (lansoprazole), - contraindication to treatment drugs,
* pregnant or lactating women,
* severe concurrent disease
* Patients who cannot give informed consent by himself or herself.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Eradication rate according to Intention to treat (ITT) and per-protocol (PP) analysis | 6 weeks
  C13-UBT will be used to assess the existence of H. pylori

SECONDARY OUTCOMES:
Incidence of adverse effects | during eradication therapy
  to assess the adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Ming Liou, MD, Principal Investigator — National Taiwan University Hospital; Ming-Shiang Wu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Romano M, Cuomo A, Gravina AG, Miranda A, Iovene MR, Tiso A, Sica M, Rocco A, Salerno R, Marmo R, Federico A, Nardone G. Empirical levofloxacin-containing versus clarithromycin-containing sequential therapy for Helicobacter pylori eradication: a randomised trial. Gut. 2010 Nov;59(11):1465-70. doi: 10.1136/gut.2010.215350. PMID 20947881
- [Derived] Liou JM, Chen CC, Chang CY, Chen MJ, Chen CC, Fang YJ, Lee JY, Yang TH, Luo JC, Wu JY, Liou TC, Chang WH, Hsu YC, Tseng CH, Chang CC, Bair MJ, Liu TY, Hsieh CF, Tsao FY, Shun CT, Lin JT, Lee YC, Wu MS; Taiwan Gastrointestinal Disease and Helicobacter Consortium. Sequential therapy for 10 days versus triple therapy for 14 days in the eradication of Helicobacter pylori in the community and hospital populations: a randomised trial. Gut. 2016 Nov;65(11):1784-1792. doi: 10.1136/gutjnl-2015-310142. Epub 2015 Sep 3. PMID 26338825